CLINICAL TRIAL: NCT04549792
Title: An Open-Label and Long-Term Extension Study to Evaluate the Efficacy and Safety of Ustekinumab in the Treatment of Patients With Ichthyoses.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-3233
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Ichthyosis
MeSH Terms: conditions — Ichthyosis | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Each subject will receive ustekinumab at Baseline (Day 0) and Months 1, 3, 5, 7, 9, and 11. During the LTE, subjects will receive injections every 8 weeks for one year: Month 13, Month 15, Month 17, Month 19, Month 21, and Month 23. Subjects will come back in for a follow-up visit at Month 25 for an end of study visit (no drug administration).

SUMMARY:
The ichthyoses are a group of lifelong genetic disorders that share characteristics of generalized skin thickening, scaling and underlying cutaneous inflammation. The vast majority are orphan disorders and are associated with extremely poor quality of life related to social ostracism from altered appearance, associated itchiness and discomfort, and functional limitations from the skin disease. Among the more common "orphan" forms of ichthyosis are autosomal recessive congenital ichthyosis (ARCI; includes lamellar ichthyosis/LI and congenital ichthyosiform erythroderma/CIE), Netherton syndrome (NS) and epidermolytic ichthyosis (EI). However, there are dozens of other syndromic and non-syndromic ichthyotic disorders as well. Therapy is time-consuming for patients or parents and is supportive, focusing on clearance of the scaling. There are no therapies based on our growing understanding of what causes the disease. We have recently found marked elevations in Th17/IL-23 pathway cytokines and chemokines in the skin of individuals with ichthyosis, most similar to the inflammatory pattern of psoriasis. While the significance of the high expression of Th17/IL-23 pathway genes across all forms of ichthyosis studied to date is unknown, the high expression of genes of the Th17/IL-23 pathway in psoriasis is thought to be causative for the disease manifestations. We propose that IL-12/IL-23 -targeting therapeutics will safely suppress the inflammation and possibly the other features of ichthyosis, improving quality of life. As a proof-of-concept study, we propose to treat children (6 years of age and higher) and adults with ichthyotic disorders with ustekinumab in an open-label trial to serially assess clinical response to and safety of ustekinumab for this group of disorders.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent; parental consent for patients under 18 years of age (plus assent for subjects age ≥ 12 and < 18).
* Subjects are at least 6 years of age or older at the time of screening.
* Before screening visit, females must be:

  * Postmenopausal, defined as

    ≥ 45 years of age with amenorrhea for at least 18 months, OR
  * ≥ 45 years of age with amenorrhea for at least 6 months and a serum FSH level > 40 IU/mL OR
  * Of childbearing potential, in which case she must satisfy at least one of the below:

Surgically sterile (has had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or

If heterosexually active, practicing a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (e.g., condoms, diaphragm, or cervical cap, with spermicidal foam, cream, film, gel or suppository), or male partner sterilization, consistent with local regulations regarding use of birth control methods for subjects participating in clinical trials, for a period of 16 weeks after the last administration of study agent,

OR

Not heterosexually active. Abstinence is allowed as an acceptable form of contraception.

Note: If a woman participant's childbearing potential changes after start of the study (e.g., a premenarchal woman experiences menarche) or if women of childbearing potential who are not heterosexually active at screening become heterosexually active, they must agree to utilize a highly effective method of birth control, as described above.

Female participants of childbearing potential (menstrual and not surgically sterile), must have a negative serum beta-human chorionic gonadotropin (ᵦ-hCG) pregnancy test at screening and a negative urine pregnancy test at Week 0 (prior to screening visit) and agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 16 weeks after the last administration of study agent.

• Male participants who are not surgically sterilized and are heterosexually active with a woman of childbearing potential, must agree to use a barrier method of contraception (e.g., condom with spermicidal foam/gel/film/cream/suppository) and to not donate sperm during the study and for 16 weeks after last receiving study agent. Note that barrier methods must also be used in all male subjects sexually active with pregnant partners for at least 16 weeks after last study agent administration.

* Subjects must have a confirmed clinical diagnosis of ichthyosis/ichthyotic disorder, and either have completed genotype or be willing to be genotyped (genotype results will not be required for entry into the study).
* Subjects must have at least moderate erythema (ISS-erythema score ≥ 2) related to his/her ichthyosis/ichthyotic disorder.
* Subjects must be clinically judged to be immunocompetent based on baseline laboratory testing (chemistry and hematology), medical history and physical examination.
* Subjects will have baseline negative QuantiFERON®-TB gold, Hepatitis B, Hepatitis C, and HIV laboratory testing.

Exclusion Criteria:

* Subjects who are unable to provide informed consent or assent (or who do not have consent from a Legally Authorized Representative if < 18 years).
* Subjects with ichthyosis vulgaris or X-linked recessive ichthyosis.
* Subjects who have a known allergy to ustekinumab or its products.
* Female subjects who are pregnant or breastfeeding, or who are considering becoming pregnant.
* Subjects who have prior biologic use targeting IL-12/IL-23 monoclonal antibody.
* Subjects who have used a systemic retinoid or systemic anti-inflammatory agent within 4 weeks prior to baseline.
* Subjects who have used topical steroid in the previous week, retinoid or keratolytic agent in the previous 24 hours.
* Subjects with active infections or recent history of serious infections, malignancies or history of malignancies, recent immunizations with live vaccines, or any severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, psychiatric, or cerebral disease, or signs or symptoms thereof
* Subjects who are under 6 years of age at the time of screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University/Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 1
  Race: White | 9
  Race: Asian | 1
  Race: Mixed | 2
Region of Enrollment [Number; unit: participants]
  United States | 13
Subtype [Count of Participants; unit: Participants]
  Harlequin Ichthyosis (HI) | 6
  Netherton Syndrome (NS) | 3
  KRT10-EI/KRT1-EI | 2
  NIPAL4-CIE | 1
  GJA-1-Erythrokeratodermia variabilis et progressiva | 1

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Total Ichthyosis Severity Score
Description: To evaluate the efficacy of ustekinumab for ichthyosis, as measured by an at least 50% reduction in severity using the Ichthyosis Severity Score (ISS) measure. The ISS measures from 0-32, with 0 being the least clinically severe and 32 being the most clinically severe.
Time Frame: 7 months after initiation of study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 13
units on a scale | -12.2 (29.9)

2. Primary Outcome: Occurence of Bacterial and Fungal Infections
Description: To evaluate the safety of ustekinumab for ichthyosis, based on occurrence of bacterial and fungal infections
Time Frame: 7 months after initiation of study drug
Measure: Number; unit: infections
Arm/Group | Open Label
Number analyzed (Participants) | 13
infections
  Superficial skin infections | 3
  Streptococcal throat infection | 2
  Onychomycosis | 1

ADVERSE EVENTS:
Time Frame: 100 weeks
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=13)
Hospitalization secondary to sepsis (Infections and infestations) | 2 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=13)
Headache (General disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 1 (1)
Broken wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
COVID-19 Infection (Infections and infestations) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Pustular psoriasis like eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Heat exhaustion (General disorders) | 1 (2)
Increased pain associated with ichthyosis (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Strep Throat Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin pustules (Skin and subcutaneous tissue disorders) | 1 (1)
Viral exanthem (Infections and infestations) | 1 (1)
Viral gastroenteritis (Infections and infestations) | 1 (1)
Viral upper respiratory infection (Skin and subcutaneous tissue disorders) | 3 (3)
Skin Infection (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT04549792/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04549792/ICF_001.pdf